CLINICAL TRIAL: NCT02557776
Title: BRCAsearch: A Population Based Prospective Study on Screening for BRCA1 and BRCA2 Germline Mutations in Patients With Newly Diagnosed Breast Cancer Treated in Southern Sweden.
Brief Title: Written Genetic Counseling and Mutation Analysis of BRCA1 and BRCA2 to Patients With Breast Cancer
Acronym: BRCAsearch
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dnr 2009/659
Record Dates: First submitted 2015-06-03; First posted 2015-09-23 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Hereditary Breast Cancer
Keywords: BRCA1; BRCA2; hereditary breast cancer; genetic counseling
MeSH Terms: conditions — Breast Cancer, Familial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genetic testing of BRCA1 and BRCA2 (Experimental): For detailes, please see "Study procedure". Women with newely diagnosed breast cancer are offered written genetic counseling and screening of mutations in BRCA1 and BRCA2.
  Interventions: Genetic: Germline genetic testing of BRCA1 and BRCA2

INTERVENTIONS:
Genetic: Germline genetic testing of BRCA1 and BRCA2

SUMMARY:
The overall purpose of the study is to evaluate a method for offering mutation analysis of BRCA1 and BRCA2 to all patients with newly diagnosed breast cancer, regardless of age at diagnosis and family history. Information about the study as well as pre-test genetic counseling will primarily be given in a written way. In addition to that, if a study participant wishes to, she can also receive pre-test telephone genetic counseling.

DETAILED DESCRIPTION:
Study population:

All patients with newly diagnosed breast cancer in southern Sweden are offered inclusion in the SCAN-B study at the time of diagnosis pre-surgery. If they consent to that, a part of the tumor is sent to a lab in Lund, Sweden, for research purposes (RNA sequencing etc.). Patients that are included in the SCAN-B study are eligible for inclusion in BRCAsearch, see inclusion and exclusion criteria.

Study procedure (summary):

1. An envelope with written information is given to the patient at the visit to the surgeon the week after surgery. This envelope contains a written genetic counseling, information about the study, an informed consent form, psychosocial questionnaires and our contact information (telephone, e-mail). The patient can contact a genetic counselor for pre-test telephone genetic counseling if she wishes to.
2. BRCA1 and BRCA2 are analyzed by full sequencing.
3. Non-carriers are informed about the test result with a letter. Mutation carriers and VUS (variants of uncertain significance) are telephoned and given a time for an appointment at the Department of Clinical Genetics within a week.
4. Psychosocial self-reported questionnaires (HAD scale, EORTC QLQ-C30, EORTC QLQ-BR23) are delivered at 3 times: At invitation to the study, one month after information about test result, and one year after information about test result.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is included in the SCAN-B study.
2. The patient is recently diagnosed with an invasive breast cancer or a ductal cancer in situ.
3. The patient has signed an informed consent form.

Exclusion Criteria:

1. The patient is unable to understand the written information in Swedish.
2. The patient's psychological state, due to chronic och temporary reasons, is such that one could suspect that information about the study or genetic testing could be substantially detrimental to the psychological well-beeing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of BRCA1/2 mutations in an unselected breast cancer cohort in southern Sweden | 3 years
Uptake of genetic testing | 3 years
Proportion of the mutation carriers that do not fulfil current criteria for genetic testing | 3 years

SECONDARY OUTCOMES:
How many of the patients that contact us for questions | 3 years
How uptake of genetic testing varies with the age at diagnosis | 3 years
  Proportion of patients tested in seperate age groups of 10 years.
The patients' attitudes towards the method used for identifying mutation carriers | 3 years
  A questionnaire with 7 general questions (answers graded 1 to 4, where 1 = not at all, and 4 = to a high extent) will be sent the participants one year after the test results were delivered. The questions are in Swedish; translated to English, examples of questions are: "are you content with the method used in the study for informtion?", "would yout have liked to have more oral information?", "are you content with having gone through genetic testing?", "would you recommend a friend of you with breast cancer to pursue genetic testing in the way that you have done?"
Psychosocial comparisons between mutation carriers and non-carriers | 4 years
  Matched comparisons between mutation carriers and non-carriers for psychosocial endpoints will be done in a nested case-control study, where two controls are selected for each mutation carrier on the basis of age, adjuvant chemotherapy, stage and ER status.

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Loman, MD, PhD, Principal Investigator — Head of Section for Breast Cancer, Melanoma and CNS tumors. Dept of Oncology, Skane University Hospital, Lund, Sweden
Locations (2):
- Sweden (2):
  - Helsingborg Hospital, Dept of Surgergy, Helsingborg
  - Kristianstad Central Hospital, Kristianstad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson MP, Torngren T, Henriksson K, Kristoffersson U, Kvist A, Silfverberg B, Borg A, Loman N. BRCAsearch: written pre-test information and BRCA1/2 germline mutation testing in unselected patients with newly diagnosed breast cancer. Breast Cancer Res Treat. 2018 Feb;168(1):117-126. doi: 10.1007/s10549-017-4584-y. Epub 2017 Nov 21. PMID 29164420